CLINICAL TRIAL: NCT04500704
Title: Almonertinib Alone Versus Almonertinib Plus Chemotherapy as First-line Treatment in Patients With Epidermal Growth Factor Receptor (EGFR) Mutation Positive With Concomitant Non-EGFR Driver Gene Mutation Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer: A Multicenter, Open-label, Randomized, Control Phase III Study (ACROSS 1)
Brief Title: Almonertinib Plus Chemotherapy as First-line Treatment in Patients With EGFR Concomitant Non-EGFR Driver Gene Mutant, Locally Advanced or Metastatic NSCLC
Acronym: ACROSS1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-LK-2020-001
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonertinib 110mg PO once daily (Active Comparator): Almonertinib 110mg PO once daily.
  Interventions: Drug: Almonertinib
- Almonertinib plus carboplatin and pemetrexed (Experimental): Almonertinib 110mg PO once daily in combination with pemetrexed (500 mg/m2) plus carboplatin (AUC=5) on Day 1 of 21day cycles (every 3 weeks) for 4-6 cycles, followed by Almonertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Interventions: Drug: Almonertinib plus carboplatin and pemetrexed

INTERVENTIONS:
Drug: Almonertinib — Almonertinib 110mg PO once daily. A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Ameile
  Arms: Almonertinib 110mg PO once daily
Drug: Almonertinib plus carboplatin and pemetrexed — Almonertinib 110mg PO once daily in combination with pemetrexed (500 mg/m2) plus carboplatin (AUC=5) on Day 1 of 21day cycles (every 3 weeks) for 4-6 cycles, followed by Almonertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Other Names: Ameile
  Arms: Almonertinib plus carboplatin and pemetrexed

SUMMARY:
This is a multicenter, randomized, controlled, phase III study.

DETAILED DESCRIPTION:
Almonertinib Alone Versus Almonertinib Plus Chemotherapy as First-line Treatment in Patients With Epidermal Growth Factor Receptor (EGFR) Mutation Positive With Concomitant Non-EGFR Driver Gene Mutation Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer: A Multicenter, Open-label, Randomized, Control Phase III Study (ACROSS 1).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures, sampling and analyses.
* Male or female, age at least 18 years.
* Pathologically confirmed locally advanced or metastatic NSCLC (e.g. this may occur systemic recurrence after prior surgery for early stage disease or patients may be newly diagnosed with stage IIIB/IV disease according to AJCC v8.0). Patients must be treatment-naïve for locally advanced or metastatic NSCLC. provided all other entry criteria are satisfied.
* Prior adjuvant, neo-adjuvant therapy and concurrent radiochemotherapy is permitted (chemotherapy, radiotherapy, investigational agents) if 6 months or more have passed since completion of therapy.
* The tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), in combination with non-EGFR driver genes mutations assessed by central testing using tumour tissue sample.
* A WHO performance status equal to 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements. If only one measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and baseline tumour assessment scans are done at least 14days afar the screening biopsy is performed.
* Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at Screening:

  1. Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
  2. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.
  3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
* Male patients should be willing to use barrier contraception (i.e., condoms).
* For inclusion in study, patient must provide a written informed consent.

Exclusion Criteria:

* Treatment with any of the following:

  1. Prior treatment with systemic anti-cancer therapy for locally advancer or metastatic NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
  2. Prior treatment with an EGFR TKI.
  3. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
  4. Radiotherapy with a limited field of radiation for palliation within 4 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
  5. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug.
* Any concurrent and/or other active malignancy that has required treatment within 2 years of first dose of study drug.
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
* Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study treatment.
* Patients who received yellow-fever vaccine or other attenuated live vaccine during pemetrexed treatment.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection. Screening for chronic conditions is not required.
* Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of Almonertinib.
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
  2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
  4. Left ventricular ejection fraction (LVEF) ≤ 40%.
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

  1. Absolute neutrophil count (ANC) <1.5×109 / L
  2. Platelet count <100×109 / L
  3. Hemoglobin <90 g/L（<9 g/dL）
  4. Alanine aminotransferase > 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
  5. Aspartate aminotransferase (AST) > 2.5 × ULN if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
  6. Total bilirubin (TBL) > 1.5 × ULN if no liver metastases or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
  7. Creatinine > 1.5 × ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 × ULN.
* Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.
* History of hypersensitivity to any active or inactive ingredient of Almonertinib, or to drugs with a similar chemical structure or class to Almonertinib.
* Patients who are allergic to pemetrexed or any other component of the preparation, carboplatin or other platinum containing compounds.
* Patients with contraindications of pemetrexed and carboplatin.
* Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
* Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
* Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From baseline, then every 6 weeks, until disease progression or discontinuation from study. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  To assess the efficacy of Almonertinib compared with Almonertinib Plus carboplatin and pemetrexed as first line therapy to EGFRm+, locally advanced or metastatic NSCLC patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Assess the anti-tumor activity: OS | Start of study drug to Survival Endpoint through study completion, an average of 3 years.
  Overall survival (OS)
Assess the anti-tumor activity: ORR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression assessed up to 24 months.
  ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression assessed up to 24 months
Assess the anti-tumor activity: DCR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. The DCR is defined as the proportion of patients with a best overall response of CR, PR, or SD assessed up to 24 months.
  Disease control rate (DCR)
Assess the anti-tumor activity: DoR | DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression assessed up to 24 months.
  Duration of response (DoR)
Assess the anti-tumor activity: DepOR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. DepOR is defined as the sum of the lengths of the longest diameters of the RECIST 1.1 target lesions up to 24 months.
  Depth of response (DepOR)
Assess the safety of Almonertinib and Almonertinib plus pemetrexed and carboplatin: Number of AEs/SAEs | Continuously throughout the study until 28 days after Termination of the treatment
  Number of adverse events (AEs)/serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Peking University International Hospital, Beijing
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No